CLINICAL TRIAL: NCT03807999
Title: Nab-Paclitaxel Plus Gemcitabine Versus Gemcitabine For The First Line Treatment of Metastatic or Locally Advanced Unresectable Adenocarcinoma of The Pancreas: A Phase II Randomized Study
Brief Title: Nab-Paclitaxel Plus Gemcitabine Versus Gemcitabine For The First Line Treatment of Pancreas Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hacettepe University (Other)
Collaborators: Celgene (Industry)
Responsible Party: Principal Investigator, Suayib Yalcin, Prof. Suayib Yalcin, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AX-PANC-SY001
Record Dates: First submitted 2019-01-08; First posted 2019-01-17 (Actual); Last update posted 2019-01-17 (Actual); Status verified 2019-01

CONDITIONS: Pancreatic Neoplasm
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — 130-nm albumin-bound paclitaxel; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nab-paclitaxel + Gemcitabine (Active Comparator): Nab-paclitaxel 125 mg/m2 as 30- to 40-minute infusion (maximum infusion time not to exceed 40 minutes) once weekly for 3 weeks followed by a week of rest. plus Gemcitabine 1000 mg/m2 as a 30- to 40-minute infusion (maximum 40 minutes) once weekly for 3 weeks followed by a week of rest.
  Interventions: Drug: Nab-paclitaxel; Drug: Gemcitabine
- Gemcitabine (Experimental): Gemcitabine 1000 mg/m2 as a 30- to 40-minute infusion (maximum 40 minutes) administered weekly for 7 weeks followed by a week of rest (8-week cycle; cycle 1 only), followed by cycles of weekly administration for 3 weeks (on days 1, 8, and 15) followed by one week of rest (4-week cycle).
  Interventions: Drug: Gemcitabine

INTERVENTIONS:
Drug: Nab-paclitaxel
  Arms: Nab-paclitaxel + Gemcitabine
Drug: Gemcitabine

SUMMARY:
This is a randomized, multicenter, phase II study of with nab-paclitaxel plus gemcitabine or gemcitabine alone for the treatment of chemotherapy-naïve patients with locally advanced or metastatic pancreatic cancer.

Arm 1: Nab-paclitaxel plus gemcitabine Arm 2: Gemcitabine alone

DETAILED DESCRIPTION:
This is a randomized, multicenter, phase II study of with nab-paclitaxel plus gemcitabine or gemcitabine alone for the treatment of chemotherapy-naïve patients with locally advanced or metastatic pancreatic cancer.

Arm 1: Nab-paclitaxel plus gemcitabine Arm 2: Gemcitabine alone

Arm 1:

Nab-paclitaxel 125 mg/m2 as 30- to 40-minute infusion (maximum infusion time not to exceed 40 minutes) once weekly for 3 weeks followed by a week of rest. plus Gemcitabine 1000 mg/m2 as a 30- to 40-minute infusion (maximum 40 minutes) once weekly for 3 weeks followed by a week of rest.

OR

Arm 2:

Gemcitabine 1000 mg/m2 as a 30- to 40-minute infusion (maximum 40 minutes) administered weekly for 7 weeks followed by a week of rest (8-week cycle; cycle 1 only), followed by cycles of weekly administration for 3 weeks (on days 1, 8, and 15) followed by one week of rest (4-week cycle).

All patients will be considered for available second-line therapies or best supportive care on the discretion of the investigators.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent.
2. Histologically or cytologically confirmed treatment-naïve metastatic or locally advanced adenocarcinoma of the pancreas not amenable to curative radiotherapy or surgery.
3. Measurable disease as defined by RECIST (ie, target lesions that can be accurately measured in at least one dimension with the longest diameter ≥ 20 mm using conventional techniques or ≥ 10 mm using spiral computed tomography [CT] scan).
4. Age ≥ 18 years.
5. ECOG Performance Status 0 or 1.
6. Adequate bone marrow function: granulocyte count ≥1500 and platelet count ≥100,000 per cubic millimeter.
7. Adequate liver function as defined by the following criteria:

   * Total serum bilirubin <2 mg/dl.
   * ALP/GGT <5 x ULN.
   * Transaminases ALT/AST ≤ 2.5 x ULN.

Exclusion Criteria:

1. Any prior systemic or investigational therapy for metastatic pancreatic cancer. Systemic therapy administered alone or in combination with radiation in the adjuvant setting is permitted if it is completed > 6 months prior to the time of study enrollment.
2. Inability to comply with study and/or follow-up procedures.
3. Presence of significant comorbidity including clinically significant cardiac disease (e.g. congestive heart failure, symptomatic coronary artery disease and cardiac arrhythmias not well controlled with medication) or myocardial infarction within the last 12 months and any other major organ failure.
4. Presence of any condition that, in the opinion of the investigator, renders the subject at high risk from treatment complications or might affect the interpretation of the results of the study.
5. Presence of central nervous system or brain metastases.
6. Life expectancy <12 weeks.
7. Pregnancy (positive pregnancy test) or lactation.
8. Prior malignancy except for adequately treated basal cell skin cancer, in situ cervical cancer, adequately treated Stage I or II cancer from which the patient is currently in complete remission, or any other form of cancer from which the patient has been disease-free for 5 years.
9. Lack of physical integrity of the upper gastrointestinal tract or malabsorption syndrome.
10. Known, existing uncontrolled coagulopathy.
11. Pre-existing sensory neuropathy > grade 1.
12. Major surgery within 4 weeks of the start of study treatment, without complete recovery.
13. Concurrent/pre-existing use of coumadin. 14. Patients older than 76 years of age.

15. Patients with active infection. 16. Patients with chronic diarrhea.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2015-02-19 (Actual); Primary Completion 2018-04-01 (Actual); Study Completion 2018-11-01 (Actual)

PRIMARY OUTCOMES:
3-months deterioration-free rate | From first dose of therapy to third month of therapy, 3 months
  EORTC QLQ-C30 (validated version for Turkish using a reduction of at least 10 points as a meaningful clinical difference) will be used to calculate "time until definitive deterioration" (TUDD) and compare patients receiving first-line Nab-Paclitaxel plus Gemcitabine versus first-line gemcitabine for metastatic or locally advanced unresectable adenocarcinoma of the pancreas. EORTC QLQ-C30 scores will be calculated every four weeks following the EORTC QLQ-C30 recommendations for calculations and scoring (EORTC QLQ- C30 published manual).

SECONDARY OUTCOMES:
Overall Survival | From first dose to death or end of the therapy, 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Suayib Yalcin, Principal Investigator — Hacettepe University

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Yalcin S, Dane F, Oksuzoglu B, Ozdemir NY, Isikdogan A, Ozkan M, Demirag GG, Coskun HS, Karabulut B, Evrensel T, Ustaoglu MA, Ozdemir F, Turna H, Yavuzsen T, Aykan F, Sevinc A, Akbulut H, Yuce D, Hayran M, Kilickap S. Quality of life study of patients with unresectable locally advanced or metastatic pancreatic adenocarcinoma treated with gemcitabine+nab-paclitaxel versus gemcitabine alone: AX-PANC-SY001, a randomized phase-2 study. BMC Cancer. 2020 Mar 30;20(1):259. doi: 10.1186/s12885-020-06758-9. PMID 32228512

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-01-07): https://cdn.clinicaltrials.gov/large-docs/99/NCT03807999/Prot_SAP_000.pdf